CLINICAL TRIAL: NCT00296439
Title: Comparison of Different Counseling Methods on Serum Phosphorus Levels in Renal Patients at Hines VA Hospital
Brief Title: Nutrition Counseling to Lower Serum Phosphorus Levels
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Edward Hines Jr. VA Hospital (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: 0034
Record Dates: First submitted 2006-02-23; First posted 2006-02-27 (Estimated); Last update posted 2006-02-27 (Estimated); Status verified 2006-02

CONDITIONS: Hemodialysis; Nutrition

INTERVENTIONS:
Behavioral: Behavior

SUMMARY:
Hemodialysis patients who receive frequent weekly nutrition counseling using motivational interviewing techniques will have lower serum phosphorus levels compared to patients receiving standard treatment.

DETAILED DESCRIPTION:
Hemodialysis patients will receive weekly nutrition counseling on how to lower their serum Phosphorus levels. Motivational interviewing techniques and strategies will be employed such as reflective listening, using affirmations, and summarizing. Average serum Phosphorus levels pre-dialysis will be compared to s.Ph post counseling. This will be compared to a group receiving nutrition counseling via standard treatment on a monthly basis.

ELIGIBILITY:
Inclusion Criteria:

* ESRD patients on dialysis with serum Ph > 5.5 mg/dL four of six labs over 6 months, mentally competent

Exclusion Criteria:

* ESRD patients on dialysis with serum Ph < 5.5 mg/dL four of six labs over 6 months, mentally incompetent

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44
Dates: Start 2006-02; Study Completion 2006-02

PRIMARY OUTCOMES:
serum Phosphorus levels

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Foley, MS, Principal Investigator — Hines VA Hospital
Locations (2):
- United States (2):
  - Edward Hines,Jr., VA Hospital, Hines, Illinois
  - Hines VA Hospital, Hines, Illinois